CLINICAL TRIAL: NCT03705195
Title: Study of Sulphonylurea Synergy With Incretins
Acronym: LOGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Ruth Cordiner, Clinical Research Fellow, Specialty Registrar Diabetes and Endocrinology, University of Dundee
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018DM01
Record Dates: First submitted 2018-07-03; First posted 2018-10-15 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gliclazide

STUDY DESIGN:
Intervention Model Description: Proof-of-Concept Physiological Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention (No Intervention): All participants in study will complete two matched clamp studies (OGTT + IGII). The first matched clamp without any intervention the second matched clamp with low dose gliclazide
- Low Dose Gliclazide (Experimental): The first 8 participants will complete the dose-ranging phase of LOGIC study. Low dose gliclazide is being used a physiological stimulus. In the dose-ranging phase, 4 participants will receive 10mg gliclazide, the remaining 4 will receive 20mg gliclazide. The allocation to 10mg or 20mg will be randomised and unblinded. The study will analyse after the first 8 participants to assess which dose produces the greatest augmentation of insulin secretion when acting synergistically with the incretin effect.
  The further 12 participants will complete the study with the identified best dose.
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Gliclazide — Low dose liquid gliclazide will be used with the second matched clamp (OGTT/IGII) in visits 4 & 5.
  Other Names: Diamicron; Zicron
  Arms: Low Dose Gliclazide

SUMMARY:
The Study of Sulphonylurea Synergy with Incretins (LOGIC) is a Proof-of-Concept Physiological study in the form of two matched isoglycaemic clamps. A matched clamp consists of an of oral glucose tolerance test followed by an isoglycaemic intravenous glucose infusion (IGII). The study will investigate whether there is synergy between a physiological sulphonylurea (SU) stimulus and the incretin effect, causing augmentation of insulin secretion in patients with type 2 diabetes mellitus (T2DM). The study will take place at The Clinical Research Centre at Ninewells Hospital in Dundee over five visits. It will evaluate 20 patients with T2DM on no diabetes therapy, or metformin monotherapy.

All participants will undergo two matched clamps. The first matched clamp will be with no intervention. The second intervention matched clamp, low-dose liquid gliclazide will be administered 1-hour prior to each test. The sulphonylurea, Gliclazide, in this this instance will be used as a physiological stimulus and will only be given on two occasions as part of the second matched clamp. The first eight participants will participate in the dose-ranging phase. They will receive either 10mg or 20mg gliclazide as a stimulus to augment the incretin effect. A further twelve participants will then be recruited to complete the study utilising the dose which caused the greatest increment in insulin secretion. LOGIC will also evaluate the cohort for effect of KCNJ11 genotype on physiological response.

DETAILED DESCRIPTION:
The Study of Sulphonylurea Synergy with Incretins (LOGIC) is a Proof-of-Concept Physiological study in the form of two matched isoglycaemic clamps. A matched clamp consists of an of oral glucose bolus test followed by an isoglycaemic intravenous glucose infusion (IGII) the next day. The study will investigate whether there is synergy between a physiological sulphonylurea (SU) stimulus and the incretin effect, causing augmentation of insulin secretion in patients with type 2 diabetes mellitus (T2DM).

The study will take place at The Clinical Research Centre at Ninewells Hospital in Dundee over five visits. It will evaluate 20 patients with T2DM on no diabetes therapy, or metformin monotherapy.

The first visit is a screening visit to ensure the participant meets inclusion and exclusion criteria, and, if so, to obtain written informed consent for study. Visits 2-5 will all occur following an overnight 10-hour fast at home. The second and third visits will make up the first matched clamp. In visit 2, the participant will undergo a 75-gram oral glucose bolus with frequent blood sampling to assess the glucose variance, insulin secretion and incretin hormone response from an oral glucose stimulus. Blood glucose level (BGL) will be sampled every 5 minutes along with hormone biochemical analysis at regular defined time points. The third visit consists of an IGII to replicate the glucose curve from the OGTT to allow measurement of incretin effect. BGL will again be sampled every 5 minutes with regular biochemical analysis of hormones.

The investigators aim to establish whether a low-dose of sulphonylurea will have a synergistic role on insulin secretion with endogenously secreted GLP-1 and GIP, therefore visits four and five will complete the same matched clamp, however, low-dose liquid gliclazide will be administered 1-hour prior to each test. The sulphonylurea, Gliclazide, in this this instance will be used as a physiological stimulus and will only be given on two occasions as part of the second matched clamp. The first eight participants will receive either 10mg or 20mg gliclazide as a stimulus to augment the incretin effect. A further twelve patients will then be recruited to complete the study utilising the dose which caused the greatest increment in insulin secretion.

The comparison of these tests will investigate the hypothesis that there is a synergistic effect between low-dose sulphonylurea and augmentation of the incretin effect on the beta cell. LOGIC will also evaluate the cohort for effect of KCNJ11 genotype on physiological response. Participants will be consented for genotyping as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 80,
* Age of Diabetes Diagnoses ≥ 35
* T2DM on no treatment or metformin monotherapy
* White British
* HbA1c ≤ 8% (64mmol/mol)
* eGFR ≥ 50ml/min-1
* ALT ≤ 2.5 x ULN
* Able to consent

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* HbA1c > 8.0% (> 64mmol/mol)
* eGFR <50ml/min-1
* ALT >2.5 x ULN
* Anaemia (Haemoglobin <12.0 g/dL for women, <13.0 g/dL for men)
* Pregnancy, lactation or a female planning to conceive within the study period
* Established pancreatic disease
* Participating in clinical phase of another interventional trial/study or have done so within the last 30 days
* Any other significant medical reason for exclusion as determined by the investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Difference in insulin secretion and incretin effect between two matched clamps (presence and absence of low dose gliclazide) | Through four study visits completed over 4 weeks
  Comparison of two matched clamps (oral glucose tolerance test + isoglycaemic intravenous glucose infusion). Matched clamp 1 - control. Matched clamp 2 - low dose gliclazide. Levels of insulin/c-peptide, incretin hormones and plasma glucose will be compared in the presence and absence of low dose gliclazide

SECONDARY OUTCOMES:
Insulin secretory response analysed by KCNJ11 Genotype (E23K, E23E, K23K) | Through four study visits completed over 4 weeks
  Difference in insulin secretory response to low dose gliclazide calculated by insulin/cpeptide levels in matched clamp(gliclazide). Differences will then be compared by participants genotype e.g. insulin secretory response for E23K, E23E, K23K variants.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan R Pearson, Study Chair — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaboe K, Knop FK, Vilsboll T, Volund A, Simonsen U, Deacon CF, Madsbad S, Holst JJ, Krarup T. KATP channel closure ameliorates the impaired insulinotropic effect of glucose-dependent insulinotropic polypeptide in patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):603-8. doi: 10.1210/jc.2008-1731. Epub 2008 Dec 2. PMID 19050053
- [Background] Gloyn AL, Pearson ER, Antcliff JF, Proks P, Bruining GJ, Slingerland AS, Howard N, Srinivasan S, Silva JM, Molnes J, Edghill EL, Frayling TM, Temple IK, Mackay D, Shield JP, Sumnik Z, van Rhijn A, Wales JK, Clark P, Gorman S, Aisenberg J, Ellard S, Njolstad PR, Ashcroft FM, Hattersley AT. Activating mutations in the gene encoding the ATP-sensitive potassium-channel subunit Kir6.2 and permanent neonatal diabetes. N Engl J Med. 2004 Apr 29;350(18):1838-49. doi: 10.1056/NEJMoa032922. PMID 15115830
- [Background] Fritsche A, Stefan N, Hardt E, Schutzenauer S, Haring H, Stumvoll M. A novel hyperglycaemic clamp for characterization of islet function in humans: assessment of three different secretagogues, maximal insulin response and reproducibility. Eur J Clin Invest. 2000 May;30(5):411-8. doi: 10.1046/j.1365-2362.2000.00649.x. PMID 10809901
- [Background] Holst JJ, Vilsboll T, Deacon CF. The incretin system and its role in type 2 diabetes mellitus. Mol Cell Endocrinol. 2009 Jan 15;297(1-2):127-36. doi: 10.1016/j.mce.2008.08.012. Epub 2008 Aug 20. PMID 18786605
- [Background] Henquin JC. Regulation of insulin secretion: a matter of phase control and amplitude modulation. Diabetologia. 2009 May;52(5):739-51. doi: 10.1007/s00125-009-1314-y. Epub 2009 Mar 14. PMID 19288076
- [Derived] Cordiner RLM, Mari A, Tura A, Pearson ER. The Impact of Low-dose Gliclazide on the Incretin Effect and Indices of Beta-cell Function. J Clin Endocrinol Metab. 2021 Jun 16;106(7):2036-2046. doi: 10.1210/clinem/dgab151. PMID 33693776